CLINICAL TRIAL: NCT03337542
Title: Real-World AR101 Market-Supporting Experience Study in Peanut-Allergic Children, Active Treatment Arm Open-Label Extension Study (RAMSES OLE)
Brief Title: AR101 Real-World Open-Label Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aimmune Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARC011
Record Dates: First submitted 2017-11-06; First posted 2017-11-09 (Actual); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Peanut Allergy
Keywords: AR101; Characterized Peanut Allergen; CPNA (Characterized Peanut Allergen); OIT (oral immunotherapy); Peanut Allergy; Peanut-Allergic Children; Desensitization; Food Allergy
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment arm description (Other): Subjects will receive maintenance dosing with AR101. Maintenance doses are provided in sachets, where each sachet contains 300 mg of peanut protein. Subjects are to ingest 300 mg orally once a day during maintenance.
  Interventions: Biological: AR101

INTERVENTIONS:
Biological: AR101 — AR101

SUMMARY:
This study is enrolling participants by invitation only. This is an open-label, safety extension study for subjects who participated in the ARC007 study.

DETAILED DESCRIPTION:
This is a Phase 3, multi-center, North American, open-label, long-term, safety extension study for eligible subjects who received AR101 therapy in the ARC007 trial (NCT03126227) and completed the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Received AR101 in study ARC007
* Completed the ARC007 study
* Use of effective birth control by sexually active female subjects of childbearing potential

Key Exclusion Criteria:

* Developed a clinically significant change in health status during the ARC007 study which in the opinion of the investigator would make the subject unsuitable for participation in this study.
* Receiving a prohibited medication or anticipated use of a prohibited medication [e.g., angiotensin-converting enzyme inhibitors, angiotensin-receptor blockers or calcium channel blockers], any monoclonal antibody, any investigational peanut immunotherapy, or any other immunomodulatory therapy.
* Currently in the build-up phase of immunotherapy for any nonfood allergen.
* Currently participating in any other interventional clinical study outside of the ARC007 study that was just completed.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 243 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director of Regulatory Affairs, Study Director — Aimmune Therapeutics
Locations (60):
- United States (55):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Medical Research of Arizona, Scottsdale, Arizona
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Jonathan Corren, M.D., Inc., Los Angeles, California
  - Allergy & Asthma Associates of Southern California, Mission Viejo, California
  - Sean N. Parker Center for Allergy Research at Stanford University - Packard-El Camino Hospital, Mountain View, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Allergy & Asthma Medical Group and Research Center, San Diego, California
  - Rady Children's Hospital, Div. Allergy & Immunology, UC San Diego, San Diego, California
  - UCSF, Benioff Children's Hospital - Allergy and Immunology, San Francisco, California
  - Allergy & Asthma Associates of Santa Clara Valley Research Center, San Jose, California
  - UCLA Medical Center, Santa Monica, Santa Monica, California
  - Bay Area Allergy, Walnut Creek, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Asthma & Allergy Associates, Colorado Springs, Colorado
  - National Jewish Health, Denver, Colorado
  - Colorado Allergy & Asthma Centers, P.C., Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Sher Allergy Specialists - Center for Cough, Largo, Florida
  - Allergy Associates of the Palm Beaches, North Palm Beach, Florida
  - Sarasota Clinical Research Windom Allergy, Asthma and Sinus, Sarasota, Florida
  - University of South Florida Asthma, Allergy, and Immunology Clinical Research Unit, Tampa, Florida
  - Atlanta Allergy & Asthma Clinic, Marietta, Georgia
  - Idaho Allergy and Research, Eagle, Idaho
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - The University of Chicago Medicine, Comer Children's Hospital, Chicago, Illinois
  - Sneeze, Wheeze, & Itch Associates, LLC, Normal, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Family Allergy & Asthma Research Institute, Louisville, Kentucky
  - Chesapeake Clinical Research, Inc., Baltimore, Maryland
  - Johns Hopkins Hospital, Pediatric Clinical Research Unit, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Division of Allergy and Clinical Immunology, Ann Arbor, Michigan
  - Clinical Research Institute, Inc., Plymouth, Minnesota
  - Children's Mercy on Broadway, Kansas City, Missouri
  - Atlantic Research Center, Ocean City, New Jersey
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Northwell Health System, Great Neck, New York
  - Univ. of Rochester Medical Center, Golisano Children's Hosp., Rochester, New York
  - University of North Carolina at Chapel Hill, Clinical & Translational Research Center, Chapel Hill, North Carolina
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Oklahoma Institute of Allergy and Asthma Clinical Research, LLC, Oklahoma City, Oklahoma
  - Columbia Asthma & Allergy Clinic, Clackamas, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - National Allergy and Asthma Research, LLC, North Charleston, South Carolina
  - Specially for Children Allergy, Asthma and Immunology Clinic, Austin, Texas
  - Children's Health, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Texas Children's Hospital, Baylor College of Medicine, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - ASTHMA Inc. Clinical Research Center, Seattle, Washington
- Canada (5):
  - McMaster University Medical Center, Hamilton, Ontario
  - Triple A Lab / Hamilton Allergy, Hamilton, Ontario
  - Cheema Research Inc. (CRI), Mississauga, Ontario
  - Ottawa Allergy Research Corp, Ottawa, Ontario
  - Gordon Sussman Clinical Research, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nilsson C, Scurlock AM, Dellon ES, Brostoff JM, Pham T, Ryan R, Brown KR, Adelman DC, Aceves SS. Onset of eosinophilic esophagitis during a clinical trial program of oral immunotherapy for peanut allergy. J Allergy Clin Immunol Pract. 2021 Dec;9(12):4496-4501. doi: 10.1016/j.jaip.2021.07.048. Epub 2021 Aug 11. No abstract available. PMID 34389504

RESULTS

PARTICIPANT FLOW:
Groups:
- AR101: Subjects will receive maintenance dosing with AR101. Maintenance doses are provided in sachets, where each sachet contains 300 mg of peanut protein. Subjects are to ingest 300 mg orally once a day during maintenance.
  AR101: AR101 powder provided in sachets
Period: Overall Study
Arm/Group | AR101
Started | 243
Safety Population | 242
Completed | 222
Not Completed | 21
Not completed — Withdrew Consent | 17
Not completed — Allergic Adverse Event | 1
Not completed — Chronic /Recurrent GI Adverse Event/Symptoms | 1
Not completed — Lost to Follow-up | 1
Not completed — Unable to Participate in Study Due to Relocation | 1

BASELINE CHARACTERISTICS:
Population: A total of 243 subjects were enrolled. However, only 242 subjects were included in Safety Population. The Safety Population is defined as all subjects who received at least 1 dose of AR101.
Arm/Group | AR101
Number analyzed (Participants) | 242
Age, Continuous [Median (Full Range); unit: years] — Age was calculated relative to the date of informed consent in ARC007
  years | 9 [4 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84
  Male | 158
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 227
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 31
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 7
  White | 174
  More than one race | 25
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (Safety and Tolerability)
Description: Number of participants with treatment-emergent adverse events including serious adverse events during the overall study period (safety and tolerability)
Time Frame: Approximately 6 months
Population: Safety population defined as all subjects who received at least 1 dose of AR101.
Measure: Count of Participants; unit: Participants
Arm/Group | AR101
Number analyzed (Participants) | 242
Participants
  Subjects with at least 1 Adverse Event (AE) | 219
  Mild AE | 176
  Moderate AE | 43
  Severe AE | 0
  Life-threatening AE | 0
  Death AE | 0
  Subjects with at least 1 Serious Adverse Event (SAE) | 1
  Mild SAE | 0
  Moderate SAE | 1
  Severe SAE | 0
  Life-threatening SAE | 0
  Death SAE | 0

2. Secondary Outcome: Number of Participants With Premature Discontinuation of Dosing Due to Adverse Events
Time Frame: Approximately 6 months
Population: Safety population defined as all subjects who received at least 1 dose of AR101
Measure: Count of Participants; unit: Participants
Groups:
- AR101: Subjects will receive maintenance dosing with AR101. Maintenance doses are provided in sachets, where each sachet contains 300 mg of peanut protein. Subjects are to ingest 300 mg orally once a day during maintenance
  AR101: AR101 powder provided in sachets
Arm/Group | AR101
Number analyzed (Participants) | 242
Participants | 1

3. Secondary Outcome: Number of Participants With Early Discontinuation of Dosing Due to Chronic/Recurrent GI Adverse Events
Time Frame: Approximately 6 months
Population: Safety population defined as all subjects who received at least 1 dose of AR101
Measure: Count of Participants; unit: Participants
Arm/Group | AR101
Number analyzed (Participants) | 242
Participants | 1

4. Secondary Outcome: Percentage of Subjects With Chronic/Recurrent GI Adverse Events Resolving Before 2, Between 2 and 4, Between 4 and 12, and ≥ 12 Weeks After Discontinuation of Dosing
Time Frame: Approximately 6 months
Population: Safety population defined as all subjects who received at least 1 dose of AR101 Number of participants analyzed: subjects who discontinued dosing due to chronic/recurrent gastrointestinal adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | AR101
Number analyzed (Participants) | 1
Participants
  < 2 weeks | 1
  2-4 weeks | 0
  4-12 weeks | 0
  ≥ 12 weeks | 0

5. Secondary Outcome: Number of Participants With Allergic Hypersensitivity Adverse Events
Time Frame: Approximately 6 months
Population: Safety population defined as all subjects who received at least 1 dose of AR101.
  Threshold of allergic hypersensitivity AE reporting ≥ 5%
Measure: Count of Participants; unit: Participants
Arm/Group | AR101
Number analyzed (Participants) | 242
Participants
  Throat irritation | 43
  Pruritus | 39
  Abdominal pain | 30
  Abdominal discomfort | 28
  Urticaria | 27
  Cough | 24
  Anaphylactic reaction | 21
  Nausea | 19
  Vomiting | 19
  Rash | 17
  Oral pruritus | 14
  Rhinorrhoea | 14

6. Secondary Outcome: Number of Participants With of Anaphylaxis as Defined in the Protocol
Description: Anaphylaxis is likely when any 1 of the 3 following sets of criteria is fulfilled:
  1. Acute onset of an illness (minutes to hours) with involvement of: (a) Skin/mucosal tissue (eg, generalized hives, itch/flush, swollen lips/tongue/uvula); AND (b) Airway compromise (eg, dyspnea, stridor, wheeze/bronchospasm, hypoxia, reduced PEFR); AND/OR (c) Reduced BP or associated symptoms (eg, hypotonia, syncope, incontinence).
  2. Two or more of the following that occur rapidly after exposure to the allergen (minutes to hours): (a) Skin/mucosal tissue; (b) Airway compromise; (c) Reduced BP or associated symptoms; (d) Persistent GI symptoms (eg, nausea, vomiting, crampy abdominal pain).
  3. Reduced BP after exposure to the allergen (minutes to hours). Infants and children: low systolic BP (age-specific) or > 30% drop in systolic BP; Adults: systolic BP < 90 mm Hg or > 30% drop from their baseline.
Time Frame: Approximately 6 months
Population: Safety population defined as all subjects who received at least 1 dose of AR101.
Measure: Count of Participants; unit: Participants
Arm/Group | AR101
Number analyzed (Participants) | 242
Participants | 21

7. Secondary Outcome: Number of Participants With Epinephrine Use as Rescue Medication
Time Frame: Approximately 6 months
Population: Safety population defined as all subjects who received at least 1 dose of AR101.
Measure: Count of Participants; unit: Participants
Arm/Group | AR101
Number analyzed (Participants) | 242
Participants | 19

8. Secondary Outcome: Number of Participants With Accidental/Nonaccidental Ingestion of Peanut and Other Allergenic Foods
Description: Number of participants with accidental/nonaccidental ingestion of peanut (not AR101 or food challenge material) and other allergenic foods.
Time Frame: Approximately 6 months
Population: Safety population defined as all subjects who received at least 1 dose of AR101.
Measure: Count of Participants; unit: Participants
Arm/Group | AR101
Number analyzed (Participants) | 242
Participants | 33

9. Secondary Outcome: Assessment of Asthma Control Using the Childhood Asthma Control Test (C-ACT) Questionnaire Total Score From Baseline, Every 4 Weeks, Early Discontinuation and Study Exit, Ages 4-11
Description: The C-ACT for subjects aged 4 to 11 years included 4 questions for the subject and 3 questions for the parent/caregiver; the total score (sum of 7 questions) ranged from 0 (worst control) to 27 (total control).
Time Frame: Baseline, Maintenance Visit 1 (Wk 4), Maintenance Visit 2 (Wk 8), Maintenance Visit 3 (Wk 12), Maintenance Visit 4 (Wk 16), Maintenance Visit 5 (Wk 20), Maintenance Visit 6 (Wk 24), Early Discontinuation (14 days after last dose), Study Exit (~6 months)
Population: Safety population defined as all subjects who received at least 1 dose of AR101.
  The C-ACT questionnaire was not completed by all subjects and/or parents/caregivers at all protocol-defined points of collection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AR101
Number analyzed (Participants) | 169
score on a scale
  Baseline: number analyzed (Participants) | 74
  Baseline | 24 (2.58)
  Maintenance Visit 1: number analyzed (Participants) | 63
  Maintenance Visit 1 | 24.4 (2.70)
  Maintenance Visit 2: number analyzed (Participants) | 47
  Maintenance Visit 2 | 25.0 (1.97)
  Maintenance Visit 3: number analyzed (Participants) | 54
  Maintenance Visit 3 | 25.0 (2.49)
  Maintenance Visit 4: number analyzed (Participants) | 52
  Maintenance Visit 4 | 25.3 (1.88)
  Maintenance Visit 5: number analyzed (Participants) | 54
  Maintenance Visit 5 | 24.8 (2.36)
  Maintenance Visit 6: number analyzed (Participants) | 53
  Maintenance Visit 6 | 24.9 (2.31)
  Early Discontinuation: number analyzed (Participants) | 5
  Early Discontinuation | 26.4 (0.89)
  Exit Visit: number analyzed (Participants) | 59
  Exit Visit | 24.2 (3.15)
  Change from Baseline to Study Exit: number analyzed (Participants) | 55
  Change from Baseline to Study Exit | 0.5 (2.94)

10. Secondary Outcome: Assessment of Asthma Control Using the Asthma Control Test (ACT) Questionnaire Total Score From Baseline, Every 4 Weeks, Early Discontinuation and Study Exit, Ages 12-17
Description: The ACT for subjects aged 12 to 17 years consisted of 5 questions, and the total score (sum of 5 questions) ranged from 5 (worst control) to 25 (total control).
Time Frame: as for outcome 9
Population: Safety population defined as all subjects who received at least 1 dose of AR101.
  The ACT questionnaire was not completed by all subjects and/or parents/caregivers at all protocol-defined points of collection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AR101
Number analyzed (Participants) | 73
score on a scale
  Baseline: number analyzed (Participants) | 42
  Baseline | 23.3 (1.92)
  Maintenance Visit 1: number analyzed (Participants) | 39
  Maintenance Visit 1 | 23.8 (1.70)
  Maintenance Visit 2: number analyzed (Participants) | 36
  Maintenance Visit 2 | 23.9 (1.65)
  Maintenance Visit 3: number analyzed (Participants) | 38
  Maintenance Visit 3 | 23.7 (2.32)
  Maintenance Visit 4: number analyzed (Participants) | 37
  Maintenance Visit 4 | 23.3 (2.72)
  Maintenance Visit 5: number analyzed (Participants) | 32
  Maintenance Visit 5 | 23.6 (2.14)
  Maintenance Visit 6: number analyzed (Participants) | 33
  Maintenance Visit 6 | 23.8 (2.19)
  Early Discontinuation: number analyzed (Participants) | 2
  Early Discontinuation | 21.5 (4.95)
  Exit Visit: number analyzed (Participants) | 35
  Exit Visit | 23.5 (2.58)
  Change from Baseline to Study Exit: number analyzed (Participants) | 35
  Change from Baseline to Study Exit | 0.3 (2.68)

11. Secondary Outcome: Number of Participants With Adverse Events That Led to Early Withdrawal
Time Frame: Approximately 6 months
Population: Safety population defined as all subjects who received at least 1 dose of AR101.
Measure: Count of Participants; unit: Participants
Arm/Group | AR101
Number analyzed (Participants) | 242
Participants | 1

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Treatment Arm Description: Subjects will receive maintenance dosing with AR101. Maintenance doses are provided in sachets, where each sachet contains 300 mg of peanut protein. Subjects are to ingest 300 mg orally once a day during maintenance.
  AR101: AR101 powder provided in sachets
Arm/Group | Treatment Arm Description
All-Cause Mortality (participants affected / at risk) | 0/242
Serious Adverse Events (participants affected / at risk) | 1/242
Other Adverse Events (participants affected / at risk) | 219/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm Description (N=242)
Anaphylactic reaction (Immune system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm Description (N=242)
Abdominal discomfort (Gastrointestinal disorders) | 45
Vomiting (Gastrointestinal disorders) | 39
Abdominal pain (Gastrointestinal disorders) | 34
Nausea (Gastrointestinal disorders) | 30
Abdominal pain upper (Gastrointestinal disorders) | 15
Oral pruritis (Gastrointestinal disorders) | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 47
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 43
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 23
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 23
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 23
Wheezing (Respiratory, thoracic and mediastinal disorders) | 17
Sneezing (Respiratory, thoracic and mediastinal disorders) | 12
Upper respiratory tract infection (Infections and infestations) | 42
Nasopharyngitis (Infections and infestations) | 19
Viral infection (Infections and infestations) | 13
Pruritus (Skin and subcutaneous tissue disorders) | 41
Urticaria (Skin and subcutaneous tissue disorders) | 33
Rash (Skin and subcutaneous tissue disorders) | 22
Pyrexia (General disorders) | 30
Headache (Nervous system disorders) | 31
Anaphylactic reaction (Immune system disorders) | 21
Eye pruritus (Eye disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Institutions cannot publish until the multi-center sponsor publication is published
* Or, institutions cannot publish until 18 months after study completion
* And Sponsor review of any publications is required prior to any institution publications according to contractual agreements

DOCUMENTS (2):
  • Study Protocol (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT03337542/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT03337542/SAP_001.pdf